CLINICAL TRIAL: NCT02277288
Title: Does Intraoperative Bladder Instillation Decrease Outpatient Recovery Time After Mid-Urethral Sling
Brief Title: Does Bladder Instillation Reduce Time to Discharge After Sling Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer T. Anger, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: Pro00026292
Record Dates: First submitted 2014-10-16; First posted 2014-10-29 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Emptied bladder arm (No Intervention): No instillation of fluid into bladder.
- Filled bladder arm (Experimental): Instilled bladder with fluid.
  Interventions: Other: Filled bladder arm

INTERVENTIONS:
Other: Filled bladder arm — Bladder to be instilled with 200 cc fluid during cystoscopy and no catheter for all mid-urethral sling procedures.
  Arms: Filled bladder arm

SUMMARY:
The purpose of this randomized control trial study is to determine if intraoperative bladder instillation of fluid decreases the time to discharge after having an outpatient mid-urethral sling procedure, and to measure the cost savings of this decrease in hospital stay. Charges will be broken down between recovery room charges and discharge area, as recovery room charges are significantly higher. The investigators suspect that a shorter time in the recovery room will translate into fewer charges.

DETAILED DESCRIPTION:
Urinary stress incontinence affects 4-35% of women. Due to the large economic impact and prevalence of the disease, urinary incontinence is a significant public health issue. With rising healthcare costs it has become increasingly important to manage patient care in the most cost-efficient manner. Considering the increasing number of women undergoing mid-urethral sling procedures, it is imperative that perioperative care is streamlined in order to minimize cost. The Cedars-Sinai Center for Continence and Women's Pelvic Health instituted a new practice pattern that enables patients to complete a voiding trial sooner after surgery compared to previous practice patterns thus allowing patients to be discharged earlier and ultimately decreasing cost. The purpose of this study is to compare the previous voiding trial practice (emptying the bladder at the end of surgery) versus the newly instituted practice (filling with bladder with 250cc) and perform a cost benefit analysis to determine if there is a significant decrease in recovery and discharge time. Both of these practices fall under the standard-of-care. However, of the several standard-of-care procedures, none have been tested for superiority. To date there are no randomized control trials that address this issue in female mid-urethral sling surgery.

Boccola et al showed in a study of 60 men who had undergone transurethral resection of the prostate (TURP) that by instilling the bladder with 300-500cc of warm saline the time to void was significantly decreased compared to standard indwelling catheter removal. It was also shown that the bladder instillation group had a significantly shorter time to discharge. The study suggested that given the significant decrease in time in recovery, this would be an ideal practice for many other outpatient procedures. Willson, et al, in another randomized trial of 75 men who underwent TURP, found that bladder infusion allowed early decision-making for discharge on the second postoperative day. Finally, McAchran and Goldman found that when patients were managed using a fast-track regimen in the outpatient setting after mid-urethral sling procedures the median time from the recovery area to discharge was less than 3 hours.

For our study, if a significant decrease in the time to discharge with the newly instituted practice pattern is demonstrated, then this practice can be adopted by other institutions and become the new standard of care to help decrease both cost and patient time in the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18 years or older
3. History of stress urinary incontinence
4. Scheduled for outpatient mid-urethral sling procedure, any approach

Exclusion Criteria:

1. Age less than 18 years
2. Pregnancy
3. Inability to give informed consent
4. History of urinary retention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time between surgery and discharge home | 2 Days
  Will analyze if the time to discharge is shorter in those patients who have had bladder instillation versus those with an indwelling catheter postoperatively.

SECONDARY OUTCOMES:
Hospital charges | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Anger, MD, MPH, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Beverly Hills, California, United States

REFERENCES:
- [Background] Boccola MA, Sharma A, Taylor C, Wong LM, Travis D, Chan S. The infusion method trial of void vs standard catheter removal in the outpatient setting: a prospective randomized trial. BJU Int. 2011 Apr;107 Suppl 3:43-6. doi: 10.1111/j.1464-410X.2011.10044.x. PMID 21492377
- [Background] Wilson ID, Bramwell SP, Hollins GW. A randomized trial comparing bladder infusion with standard catheter removal after transurethral resection of the prostate. BJU Int. 2000 Dec;86(9):993-5. doi: 10.1046/j.1464-410x.2000.00963.x. PMID 11119091
- [Background] McAchran SE, Goldman HB. Contemporary length of stay and resource utilization when using a fast-track regimen for mid-urethral sling surgery. Urology. 2009 Sep;74(3):531-4. doi: 10.1016/j.urology.2009.04.039. Epub 2009 Jul 9. PMID 19592077
- [Background] Luber KM. The definition, prevalence, and risk factors for stress urinary incontinence. Rev Urol. 2004;6 Suppl 3(Suppl 3):S3-9. PMID 16985863
- [Background] Wilson L, Brown JS, Shin GP, Luc KO, Subak LL. Annual direct cost of urinary incontinence. Obstet Gynecol. 2001 Sep;98(3):398-406. doi: 10.1016/s0029-7844(01)01464-8. PMID 11530119